CLINICAL TRIAL: NCT06619028
Title: Effectiveness of the Use of External Body Weight in the Regulation of Body Weight, Body Composition and Analytical Parameters in Adults With Grade II and III Obesity
Brief Title: External Body Weight Effects on Body Weight in Adults With Grade II and III Obesity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Escoles Universitaries Gimbernat (Other)
Collaborators: Corporacion Parc Tauli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: G0001
Record Dates: First submitted 2024-09-13; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Obesity Prevention; Obesity
Keywords: Obesity; Body Weight; Weight loss; Treatment; Leptin; Gravitostat
MeSH Terms: conditions — Obesity; Body Weight; Weight Loss

STUDY DESIGN:
Intervention Model Description: A prospective longitudinal controlled design on the use of external body weight (where patients are their own control: intrasubject controlled study) for 4 weeks, with a 4-week pre-control period and a 4-week follow-up.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (IG) (Experimental): During the intervention period, the participants will be exposed to an external load, by means of a weighted vest of 10% of their body weight, for a minimum of 8 hours per day for 4 weeks. In the first phase of the study, participants will be followed without changes in their lifestyle as a control. During the intervention they will be instructed to perform their usual activities with the vest, without further alterations in their lifestyle. This will be followed by a 4-week follow-up period without the use of the weighted vest.
  Interventions: Device: Weighted vest

INTERVENTIONS:
Device: Weighted vest — During the intervention period, the participants will be exposed to an external load, by means of a weighted vest of 10% of their body weight, for a minimum of 8 hours per day for 4 weeks. In the first phase of the study, participants will be followed without changes in their lifestyle as a control. During the intervention they will be instructed to perform their usual activities with the vest, without further alterations in their lifestyle. This will be followed by a 4-week follow-up period without the use of the weighted vest.
  Other Names: External load

SUMMARY:
Obesity is a growing problem in industrialized societies. This condition is associated with an increase in metabolic and cardiovascular diseases. Its cause is multifactorial, influenced by the environment, excessive calorie consumption, insufficient physical activity, sedentary lifestyle and alterations in energy metabolism.

In this context, the hormone leptin, responsible for regulating appetite and body weight, presents resistance in people with obesity, altering the metabolic balance. Recent research has explored the concept of the "gravitostat", a system that responds to the mechanical stimulus of standing upright, as a promising approach in the regulation of body weight. Animal and human studies have shown positive results in weight loss and body recomposition using this system. However, more research is needed to evaluate the clinical applicability and effectiveness of the gravitostat in the management of obesity.

For this reason, the present study is proposed, with a prospective longitudinal controlled design in the use of external body weight (where the patients are their own control: intrasubject controlled study) during 4 weeks, with a previous control period of 4 weeks and a follow-up of 4 weeks. The proposed objectives are to analyze the effectiveness of the use of external weight in the regulation of body weight, body composition and analytical parameters in people with grade II and III obesity. In this way, to analyze the clinical applicability of the gravitostat in the management of patients with this metabolic pathology.

DETAILED DESCRIPTION:
BACKGROUND Obesity is one of the most prevalent and booming health and social problems in recent decades in industrialized societies. Obesity rates in European countries such as the United Kingdom, Germany, France and Spain fluctuate between 23 and 29% in the adult population, according to the World Health Organization (WHO). These values increase to 42.4%, 27% and 31% in the United States, Canada and Australia, respectively, considering data from the last 5 years from the main health agencies of these countries, making it a social and public health problem.

The etiopathogenesis of this condition is multifactorial; the obesogenic characteristics of the environment can influence gene expression conditioning the development of obesity. Increased caloric intake, influenced by high-fat diets (Westerns' diet), the absence or insufficiency of physical activity and alterations in energy metabolism seem to be the three fundamental factors contributing to the development of obesity. Moreover, these factors seem to play a major role in the development of other metabolic entities such as hypertension, dyslipidemia and insulin resistance or type II diabetes, which, together with central obesity, make up the metabolic syndrome. This clinical entity doubles the risk of coronary and cerebrovascular disease, increases the risk of diabetes fivefold, and increases all-cause mortality by 50%. In parallel to the risk factors listed above, some studies highlight the role of a sedentary lifestyle as a factor independent of physical activity in contributing to the development of metabolic pathology. Not only the absence of low, moderate or high intensity physical activity has been correlated with the development of metabolic syndrome, but also the increase in time spent in sedentary activities, with an odds ratio of 2.38.

These intrinsic and extrinsic factors seem to interact and condition each other, altering homeostatic and physiological processes in obese individuals.

Since its discovery and description in the 1990s by Friedman leptin has been the most important hormonal factor in the regulation and control of caloric intake and metabolism, and consequently of body weight and composition. Its peripheral production at the level of white fat tissue and its hypothalamic effects (decrease in orexic neuronal activity and conditioning of dopaminergic reward circuits) condition the individual's response to food, regulating satiety and intake.

Evidence shows that this mechanism is altered in people with obesity where excessive leptin production, due to increased concentrations of fat tissue, and consequently high serum concentrations, condition central and peripheral sensitivity to this hormone, generating, in the long run, lower response efficiency, giving rise to the term "leptin resistance ". This resistance seems to modify the hypothalamic satiety signal, as well as the dopaminergic circuits associated with food intake,predisposing to the appearance or increase of metabolic pathology, especially obesity. This dysregulation in caloric intake appears without alterations in the production and function of ghrelin, a hormone produced in the stomach associated with hunger.

Recent research has proposed a second system of body weight homeostasis associated with the mechanical stimulus of standing upright, coined the term "gravitostat ".

Studies in mice and in humans show promising results in the regulation of body weight and fat percentage by this mechanical system. These investigations have shown significant reductions in both parameters when external weight is added to the study subjects, generating modifications in food intake and caloric expenditure. These adaptations have been tested independently of leptin resistance or the lack of leptin receptors, thus demonstrating the existence of an independent homeostatic regulation pathway. These changes have been shown to be significant only in obese subjects, whereas in normopese subjects, who show greater sensitivity to leptin, the changes produced by the increased load do not appear to be significant. Regarding body recomposition, these studies seem to indicate a maintenance of muscle mass, without experiencing significant losses, as in other contexts of caloric deficit thus prioritizing the loss of white fat tissue (especially visceral) as a mechanism of weight regulation.

Some studies justify this action by the production of fibroblast growth factors (FGF) produced by the osteocytes, specifically, the factor FGF21 associated with the hypothalamic receptor FGFR1c. The triplication in the serum quantities of FGF21 factor, by hepatic expression, in subjects exposed to body weight, seems to justify the increase in fat mobilization and oxidation, as well as the loss of body weight, which, despite the catabolic context, does not affect muscle mass. In any case, the results do not yet seem to be conclusive, since at supraphysiological loads of FGF21 the action of weight loss is mitigated, probably indicating a regulation by the FGFR1c receptor mediated, in part, by one or more other factors. This could be a key factor in the lack of effectiveness in normopese individuals.

Some stuides show how the increased load during the prepubertal period in rats reduces the expression of hormones associated with growth (IGF-1 and GHGH) as a homeostatic mechanism to control sudden weight gain. Similarly, down-regulation of ghrelin receptors at the hypothalamic level is observed, leading to a decrease in caloric intake. Other adaptations that could explain the physiological mechanism of body homeostasis, in this case, during growth.

With respect to analytical parameters, the only clinical trial carried out in humans only shows significant reductions in LDL and leptin; the results are inconclusive for the other parameters studied.

Taking this into consideration, some evidence observed a bidirectional regulation, with increases in body weight and fat mass in subjects with the sudden decrease in load. The lack of follow-up in human studies4 does not allow extrapolation of these results. At the clinical level, this regulation could justify weight and, essentially, fat gain after liposuction interventions6 or other contexts of abrupt weight loss or dietary patterns with aggressive caloric restriction. In this case, both homeostatic systems would influence, on the one hand, the gravitostat would increase food intake and the decrease in adipose tissue and the conditioned reduction in leptin production would decrease anorexic signals, predisposing the subjects to have more frequent and calorically dense intakes.

The results presented by some reserchers are promising in the development of new tools to help patients with obesity, despite this, the short duration of the intervention and the lack of follow-up of the patients, the lack of consistent changes in the analytical analysis, the performance only in young and moderately obese patients, as well as the high demand of the intervention protocol and the sudden gain in body weight after the intervention (in basic studies) make further research necessary to prove the applicability, usefulness and effectiveness of the gravitostat as a therapeutic tool, as well as the high demands of the intervention protocol and the sudden gain of body weight after the intervention (in basic studies) make it necessary to carry out further research to prove the applicability, usefulness and effectiveness of the gravitostat as a therapeutic tool in patients with obesity.

For this reason, the present doctoral thesis proposes an intrasubject controlled study for a period of 12 weeks (4 control, 4 intervention and 4 follow-up) in patients with grade II and III obesity. During the intervention period, the participants will be exposed to an external load, by means of a weighted vest of 10% of their body weight, for a minimum of 8 hours per day for 4 weeks. In the first phase of the study, participants will be followed without changes in their lifestyle as a control. During the intervention, they will be instructed to perform their usual activities with the vest, without further alterations in their lifestyle.

For this study, accepting an alpha risk of 0.05 and a beta risk of less than 0.2 in a unilateral contrast, 24 patients are required to detect a difference equal to or greater than 0.15 unit. A common standard deviation of 1.4 and a correlation between the first and second measurement of 0.99 (according to literature) is assumed. A loss rate of 10% is assumed. Patients will be recruited from the endocrinology service of the Hospital Universitario Parc Taulí.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* BMI (≥35)
* Compliance at intervention delivery.

Exclusion Criteria:

* Chronic pathology that may hinder the performance of the intervention
* Chronic pain
* Regular consumption of pharmacology or supplementation that affects body weight
* Inability to perform any physical activity or high risk of suffering adverse effects from the interventibariatric-metabolic surgery
* Reduced mobility
* Changes of 5kg or more in the last 3 months
* Drastic changes in lifestyle habits in the last 3 months (physical activity, eating habits, nicotine or alcohol consumption)
* Apparent risk of not being able to complete the study intervention (at the principal investigator's discretion)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Body weight | From enrollment to the end of treatment at 12 weeks
  Measured fasting weight by electronic scale (BC-545N Tanita)

SECONDARY OUTCOMES:
Nutritional state | From enrollment to the end of treatment at 12 weeks
  Short Dietary Questionnaire Punctuation: From 0 to 9. Interpretation: Higher results, better adherence with Mediterranean diet. Lower results, worst adherence with Mediterranean diet.
Grip Strength | From enrollment to the end of treatment at 12 weeks
  Measuring tool: Grip Strength Dynamometer Takei T.K.K 5401 Procedure: 3 consecutive measurements with each extremity, taking the mean as reference value for each.
Lower Extremity Strength | From enrollment to the end of treatment at 12 weeks
  30' chair stand-up test Test performed only once, with a 43 cm (17 inches) high chair without armrests.
Activity state | From enrollment to the end of treatment at 12 weeks
  Minnesota Leisure Time Physical Activity Questionnaire No standared punctuation Higher values associated with higher activity state Punctuation registred in minutes, days, months.
Absolute frequency of patients reporting adverse effects | From week 4 to the end of treatment at 12 weeks
  Self-reported ad hoc questionnaire following CTCAE v4.0 criteria
Body compostiton | From enrollment to the end of treatment at 12 weeks
  Bioimpedance electrical analysis (BC-545N Tanita) Body fat percentage; no standarized values, lower values are better. Muscle mass percentatge; no standarized values, higher values are better. Bone mass level; no standarized values, higher values are better. Visceral fat level; no standarized values, lower values are better.
Body compostiton | From enrollment to the end of treatment at 12 weeks
  Ultrasound measurement of muscle cross-sectional area and fat folds in thigh and abdomen (General Electric VScan) Muscle cross-sectional area: mesured (midpoint from anterosuperior iliac spine and superior pole of patella). 3 mesurements, mean result.
  Fat fold: mesured (midpoint from anterosuperior iliac spine and superior pole of patella). 3 mesurements, mean result.
  Fat fold: mesured (2cm below the umbilicus; subumbilical area). 3 mesurements, mean result.
Age | Baseline
  Measured in ages using a self-reported questionnaire.
Sex | Baseline
  Measured in dichotomous variable using a self-reported questionnaire.
Height | Baseline
  Measurement in centimeters using tape measure
Body Mass Index | Baseline
  Calculated by height in meters and weight in kilograms. Following this formula: BMI = weight ÷ height^2 (units: kg/m^2)
  Fallowing this criteria to interpret:
  * lt; 16.0 Severely Underweight 16.0 - 18.4 Underweight 18.5 - 24.9 Normal 25.0 - 29.9 Overweight 30.0 - 34.9 Type I Obesity 35.0 - 39.9 Type II Obesity
  * gt; 40.0 Type III Obesity

CONTACTS AND LOCATIONS:
Overall Officials: Maria Assumpta Caixàs Pedragós, PhD, MD, Principal Investigator — Consorci Sanitari Parc Taulí
Locations (1):
- EUGimbernat, Sant Cugat del Vallès, Barcelona, Spain

REFERENCES:
- [Result] Palsdottir V, Windahl SH, Hagg DA, Keantar H, Bellman J, Buchanan A, Vaughan TJ, Linden D, Jansson JO, Ohlsson C. Interactions Between the Gravitostat and the Fibroblast Growth Factor System for the Regulation of Body Weight. Endocrinology. 2019 May 1;160(5):1057-1064. doi: 10.1210/en.2018-01002. PMID 30888399
- [Result] Bake T, Peris-Sampedro F, Waczek Z, Ohlsson C, Palsdottir V, Jansson JO, Dickson SL. The gravitostat protects diet-induced obese rats against fat accumulation and weight gain. J Neuroendocrinol. 2021 Aug;33(8):e12997. doi: 10.1111/jne.12997. Epub 2021 Jul 9. PMID 34240761
- [Result] Jansson JO, Dalmau Gasull A, Schele E, Dickson SL, Palsdottir V, Palmquist A, Girones FF, Bellman J, Anesten F, Hagg D, Ohlsson C. A Body Weight Sensor Regulates Prepubertal Growth via the Somatotropic Axis in Male Rats. Endocrinology. 2021 Jun 1;162(6):bqab053. doi: 10.1210/endocr/bqab053. PMID 33693673
- [Result] Jansson JO, Palsdottir V, Hagg DA, Schele E, Dickson SL, Anesten F, Bake T, Montelius M, Bellman J, Johansson ME, Cone RD, Drucker DJ, Wu J, Aleksic B, Tornqvist AE, Sjogren K, Gustafsson JA, Windahl SH, Ohlsson C. Body weight homeostat that regulates fat mass independently of leptin in rats and mice. Proc Natl Acad Sci U S A. 2018 Jan 9;115(2):427-432. doi: 10.1073/pnas.1715687114. Epub 2017 Dec 26. PMID 29279372
- [Result] Ohlsson C, Hagg DA, Hammarhjelm F, Dalmau Gasull A, Bellman J, Windahl SH, Palsdottir V, Jansson JO. The Gravitostat Regulates Fat Mass in Obese Male Mice While Leptin Regulates Fat Mass in Lean Male Mice. Endocrinology. 2018 Jul 1;159(7):2676-2682. doi: 10.1210/en.2018-00307. PMID 29800288
- [Result] Ohlsson C, Gidestrand E, Bellman J, Larsson C, Palsdottir V, Hagg D, Jansson PA, Jansson JO. Increased weight loading reduces body weight and body fat in obese subjects - A proof of concept randomized clinical trial. EClinicalMedicine. 2020 Apr 30;22:100338. doi: 10.1016/j.eclinm.2020.100338. eCollection 2020 May. PMID 32510046
- [Result] Ekblom O, Ekblom-Bak E, Rosengren A, Hallsten M, Bergstrom G, Borjesson M. Cardiorespiratory Fitness, Sedentary Behaviour and Physical Activity Are Independently Associated with the Metabolic Syndrome, Results from the SCAPIS Pilot Study. PLoS One. 2015 Jun 29;10(6):e0131586. doi: 10.1371/journal.pone.0131586. eCollection 2015. PMID 26120842
- [Result] Gallardo-Alfaro L, Bibiloni MDM, Mascaro CM, Montemayor S, Ruiz-Canela M, Salas-Salvado J, Corella D, Fito M, Romaguera D, Vioque J, Alonso-Gomez AM, Warnberg J, Martinez JA, Serra-Majem L, Estruch R, Fernandez-Garcia JC, Lapetra J, Pinto X, Garcia Rios A, Bueno-Cavanillas A, Gaforio JJ, Matia-Martin P, Daimiel L, Mico-Perez RM, Vidal J, Vazquez C, Ros E, Fernandez-Lazaro CI, Becerra-Tomas N, Gimenez-Alba IM, Zomeno MD, Konieczna J, Compan-Gabucio L, Tojal-Sierra L, Perez-Lopez J, Zulet MA, Casanas-Quintana T, Castro-Barquero S, Gomez-Perez AM, Santos-Lozano JM, Galera A, Basterra-Gortari FJ, Basora J, Saiz C, Perez-Vega KA, Galmes-Panades AM, Tercero-Macia C, Sorto-Sanchez C, Sayon-Orea C, Garcia-Gavilan J, Munoz-Martinez J, Tur JA. Leisure-Time Physical Activity, Sedentary Behaviour and Diet Quality are Associated with Metabolic Syndrome Severity: The PREDIMED-Plus Study. Nutrients. 2020 Apr 7;12(4):1013. doi: 10.3390/nu12041013. PMID 32272653
- [Result] Berthoud HR, Morrison CD, Munzberg H. The obesity epidemic in the face of homeostatic body weight regulation: What went wrong and how can it be fixed? Physiol Behav. 2020 Aug 1;222:112959. doi: 10.1016/j.physbeh.2020.112959. Epub 2020 May 16. PMID 32422162